CLINICAL TRIAL: NCT07299487
Title: Evaluation of a Diagnostic Aid Tool for the Management of Vertigo Patients for General Practitioners : A Retrospective, Single-center Study at the Strasbourg University Hospital.
Brief Title: Diagnostic Aid for Vertigo Patients
Acronym: ADPV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9374
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Vertigo
Keywords: Vertigo
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Consultations for vertigo in general practice are difficult, primarily due to practitioners' lack of experience. Patient referrals can be inaccurate, leading to missed opportunities or misuse of resources. The creation of a diagnostic aid flowchart that provides referrals will improve patient care and reassure general practitioners during consultations for vertigo.

ELIGIBILITY:
Inclusion Criteria:

* Subject of legal age (≥18 years)
* Having received initial care from a medical student and whose consultation data, interview, clinical examination, and diagnosis according to our decision tree were present in the patient file.
* Patient for whom a definitive diagnosis was made by the on-call ENT physician during the same hospital visit.

Exclusion Criteria:

* Subject who expressed objection to the reuse of their data for scientific research.
* Known chronic vestibular pathology
* Incomplete patient medical file
* Patient examined outside the ENT department.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject having received initial care from a medical student and whose consultation data, interview, clinical examination, and diagnosis according to our decision tree were present in the patient file.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of concordance between the diagnosis in the decision tree and the diagnosis made by an ENT (otolaryngologist) physician. | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-faciale - CHU de Strasbourg - France, Strasbourg, France